CLINICAL TRIAL: NCT02128711
Title: Mapping Chemical and Microbiological Heterogeneity Throughout Explanted Cystic Fibrosis Lung Specimens
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: PACCS-2018-27376; 4R00HL114862-02 (NIH)
Record Dates: First submitted 2014-04-25; First posted 2014-05-01 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Cystic Fibrosis
Keywords: lung; cystic fibrosis; bacteria; positive diagnosis of CF,
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Explanted lung specimens from cystic fibrosis patients. This tissue, that would otherwise be discarded, is being retained for microbiological analysis.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
There is plenty of evidence to suggest that the lung is not uniform. The internal surface area is 30 times that of skin, and the different bronchioles/bronchi/alveoli differ greatly in blood perfusion, temperature, oxygen tension, and pH. Also, particularly in the context of respiratory disease, notable differences are present in the structure of epithelial cells, cilia, production of mucus, and inflammatory/immune responses. All of these factors are known to impact the physiology of bacteria, yet, there is very little understanding of how they impact a) the presence/absence of particular bacterial species throughout the respiratory tract, or b) the metabolic processes used by these bacteria within the human host environment. A greater understanding of the relationships between environmental (chemical) gradients in the lungs of diseased patients (particularly those with cystic fibrosis) and the microbial communities that are present may lead to novel hypotheses about manipulation of the respiratory environment for therapeutic benefit. To investigate this further, the investigators propose to use explanted lung specimens from cystic fibrosis patients to test the following hypothesis:

Hypothesis: In patients with cystic fibrosis, bacterial community composition, metabolism and environmental chemistry will vary depending on their spatial location within the airways.

DETAILED DESCRIPTION:
To study this in greater detail, the investigators propose to study explanted tissue of CF patients that are scheduled to undergo single or double lung transplant surgery as a late-stage disease therapeutic strategy. This population will be limited to the Adult CF clinic, as pediatric subjects are rarely candidates for lung transplantation. The Adult CF Clinic performs upwards of 20 surgeries per year, and tissue that is explanted is typically discarded. Using this tissue, the investigators propose the following objectives:

1. Use 16S culture-independent sequencing to characterize the spatial distribution of bacterial pathogens throughout the lungs of cystic fibrosis patients. Lungs will be dissected into 5 separate lobes, and mucus material will be collected, homogenized, and processed for bacterial species identification.
2. Perform detailed analysis of specific gene expression throughout the respiratory tract that will serve as a proxy of environmental conditions found there. Using the same approach in Aim 1, bacterial mRNA will be extracted using established procedures. A subset of environmentally-specific genes will be detected to provide a readout of bacterial metabolism in use within the CF lung environment.
3. Use in situ hybridization imaging to visualize the spatial distribution of specific bacteria and their gene expression profiles (informed by data generated in objectives 1 and 2). The bacteria and gene candidates identified/studied in Aims 1 and Aims 2 will then be subject to analysis using in situ hybridization imaging. Tissue will be processed using microtomy and fluorescent probes will be applied to image the spatial distribution of specific bacterial species and their metabolisms throughout the respiratory tract.

Information collected in these three objectives will then be paired with patient data (age, genotype, prior medical treatments, clinical microbiology data) to generate better working models of late-stage disease in CF patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of cystic fibrosis
* eligible for lung transplantation
* exhausted other available therapies without success
* informed consent

Exclusion Criteria:

* there are no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will include those undergoing single or double lung transplantation as part of their normally scheduled therapy for cystic fibrosis disease.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Composition of bacterial communities throughout an explanted lung | Entire study (3 years)
  16S culture-independent sequencing will be used to characterize the spatial distribution of bacterial pathogens throughout the lungs of cystic fibrosis patients. Explanted lung specimens will be dissected into 5 separate lobes, and mucus material will be collected, homogenized, and processed for bacterial species identification.

SECONDARY OUTCOMES:
Levels of bacterial gene expression | Entire study (3 years).
  Gene expression analysis will be used to study bacterial physiology within explanted lungs and will serve as a proxy of environmental conditions found there. Using the same approach in as outcome 1, bacterial mRNA will be extracted using established procedures. A subset of environmentally specific genes will be detected to provide a readout of bacterial metabolism in use within the CF lung environment.

OTHER OUTCOMES:
Distribution of bacterial gene expression | Entire study (3 years)
  The bacteria and their gene candidates identified in outcomes 1 and 2, will then be subject to analysis using in situ imaging. Tissue will be process using microtomy and fluorescent probes will be applied to image the spatial distribution of specific bacterial species and their metabolisms throughout the respiratory tract.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan C Hunter, PhD, Principal Investigator — University of Minnesota Medical School (Microbiology)
Locations (1):
- University of Minnesota Medical School, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Hunter RC, Asfour F, Dingemans J, Osuna BL, Samad T, Malfroot A, Cornelis P, Newman DK. Ferrous iron is a significant component of bioavailable iron in cystic fibrosis airways. mBio. 2013 Aug 20;4(4):e00557-13. doi: 10.1128/mBio.00557-13. PMID 23963183
- [Background] Hunter RC, Klepac-Ceraj V, Lorenzi MM, Grotzinger H, Martin TR, Newman DK. Phenazine content in the cystic fibrosis respiratory tract negatively correlates with lung function and microbial complexity. Am J Respir Cell Mol Biol. 2012 Dec;47(6):738-45. doi: 10.1165/rcmb.2012-0088OC. Epub 2012 Aug 3. PMID 22865623 (Retraction: PMID 30592444 Am J Respir Cell Mol Biol. 2019 Jan;60(1):134)